CLINICAL TRIAL: NCT00356083
Title: Opioid Switching From Oral Slow Release Morphine to Oral Methadone May Improve Pain Control in Chronic Non-malignant Pain: a Nine-month Follow-up Study.
Brief Title: Opioid Rotation From Morphine to Methadone in Treatment of Non-malignant Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 188-03REK
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Non-malignant Chronic Pain
MeSH Terms: interventions — Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- switch from morphine to methadon (Experimental)
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Methadone

SUMMARY:
Patients with non-malignant pain are switched from morphine to methadone with a nine-months' follow-up.

DETAILED DESCRIPTION:
Twelve patients with poor pain control or unacceptable side effects during treatment with morphine were switched to methadone and followed for nine months in this open prospective study. Primary outcomes were patient preference for opioid and pain control while physical, cognitive and role functioning were secondary outcomes. The morphine dose was decreased by 1/3 daily and was replaced with an equianalgesic dose of methadone over a three-day period. During switching and a one-week dose titration period, patients were given additional methadone if required. During dose titration one patient experienced sedation requiring naloxone. Four patients were switched back to morphine due to poor pain control, drowsiness or sweating. Seven patients preferred long-term (>nine months) treatment with methadone and reported reduced pain and improved functioning while cognition was not improved. This study brings novel information on the long-term consequences for pain control, health-related quality of life and cognitive functioning with a switch from morphine to methadone in the treatment of chronic non-malignant pain.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age
* non-malignant chronic pain
* morphine use

Exclusion Criteria:

* addiction
* kidney disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-01; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
pain | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Petter C. Borchgrevink, PhD MD, Principal Investigator — Norwegian University of Science and Technology; Petter C Borchgrevink, MD PhD, Study Chair — Norwegian University of Science and Technology

REFERENCES:
- [Background] Fredheim OM, Borchgrevink PC, Hegrenaes L, Kaasa S, Dale O, Klepstad P. Opioid switching from morphine to methadone causes a minor but not clinically significant increase in QTc time: A prospective 9-month follow-up study. J Pain Symptom Manage. 2006 Aug;32(2):180-5. doi: 10.1016/j.jpainsymman.2006.02.010. PMID 16877186
- [Result] Fredheim OM, Kaasa S, Dale O, Klepstad P, Landro NI, Borchgrevink PC. Opioid switching from oral slow release morphine to oral methadone may improve pain control in chronic non-malignant pain: a nine-month follow-up study. Palliat Med. 2006 Jan;20(1):35-41. doi: 10.1191/0269216306pm1099oa. PMID 16482756